Clinical Trial Number: NCT04731233

**Title:** A Randomized, Double-Blind Study of the Efficacy of Platelet-Rich Growth Factor (PRGF) Supplementation Compared to Steroid Supplementation After Temporomandibular Joint (TMJ) Arthrocentesis in Female Patients With TMJ Osteoarthritis (OA)

Date: January 2, 2025

**Proposed Statistical Analyses** 

## **Statistical Analyses**

Statistical analyses will consist of descriptive statistics (mean, standard deviation for parametric data; median and range for non-parametric data) and inferential statistics (two way ANOVA, 1 between (treatment groups), 1 within (time)) using a probability level of < 0.05). The primary outcome variable will be intracapsular pain.